CLINICAL TRIAL: NCT05115604
Title: Insomnia in the Patient With Schizophrenic Disorder: Evaluation of a Cognitive Behavioural and Psychoeducational Intervention
Brief Title: Insomnia in the Patient With Schizophrenic Disorder: Evaluation of a CBT and Psychoeducational Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Batalla-Martin (Other)
Responsible Party: Sponsor-Investigator, David Batalla-Martin, Principal Investigator, Nou Barris Mental Health Center
Organization: Nou Barris Mental Health Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NBMH01/2021
Record Dates: First submitted 2021-10-20; First posted 2021-11-10 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Insomnia; Schizophrenia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrervention group (Experimental): One and a half hour sessions (6 sessions) of cognitive behavioural therapy and psychoeducation. The sessions will consist of: sleep hygiene, cognitive therapy, bedtime restriction, stimulus control and relaxation.
  Interventions: Behavioral: cognitive behavioural intervention
- Control group (No Intervention): routine clinical follow-up

INTERVENTIONS:
Behavioral: cognitive behavioural intervention — Six sessions of cognitive behavioural and psychoeducational therapy will be conducted to treat insomnia.
  Arms: Intrervention group

SUMMARY:
The study aims to evaluate the efficacy of a cognitive behavioural and psychoeducational intervention in patients with insomnia and diagnosed with a schizophrenic disorder.

DETAILED DESCRIPTION:
Patients will be recruited by consecutive non-probabilistic sampling at the Outpatient Mental Health Centre of Nou Barris in Barcelona and subsequently randomised into 2 groups, control and intervention. Presence and severity of insomnia will be assessed through the following measurement instruments: ISI for presence and severity, PSQI for sleep quality and EQ-5D for health-related quality of life. Patients in intervention will attend 6 group sessions with cognitive behavioural and psychoeducational intervention and the control group will carry out the usual follow-up. Pre-post, 6-month and 9-month assessments will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia disorder (ISI scale)
* Schizophrenic disorder

Exclusion Criteria:

* Presence of severe psychopathological alteration
* Inability to understand the Spanish language or difficulties writing or reading

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2022-07-09 (Actual)

PRIMARY OUTCOMES:
Change in the severity of insomnia, mesured with the Spanish version of the Insomnia Severity Insomnia | Changes in baseline scores at 6 weeks (end of six sessions CBT - Intervention group), at 6 months (Intervention gruop & control group) and at 9 months (Intervention gruop & control group)
  Insomnia severity was assessed using the Insomnia Severity Index (ISI) (Morin, 1993), a self-applied instrument designed to briefly assess the severity of insomnia in the general population based on the diagnostic criteria of the DSM-IV and the ICSD. A 5-point Likert scale is used to rate each item (0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: not clinically significant insomnia (0-7); subthreshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28) This scale has been found to have adequate psychometric properties in studies conducted using English version (Bastien et al, 2001), with internal reliability values (Cronbach's a) between 0.74 and 0.90, and test-retest reliability equal to 0.89 one month after evaluation, 0.77 two months after, and 0.73 three months after. Two validation studies of the Spanish version of the ISI (Fernandez-Mendoza et al., 2012; Sierra et al, 2008)
Change in the quality of sleep, mesured with the Spanish version of The Pittsburgh Sleep Quality Index | Changes in baseline scores at 6 weeks (end of six sessions CBT - Intervention group), at 6 months (Intervention gruop & control group) and at 9 months (Intervention gruop & control group)
  The quality of sleep has been analysed by The Pittsburgh Sleep Quality Index, which is made up of 19 self-administered questions. The 19 self-rated questions assess a wide variety of factors relating to sleep quality, including estimates of sleep duration and latency and of the frequency and severity of specific sleep-related problems. These I9 items are grouped into seven component scores, each weighted equally on a O-3 scale. The seven component scores are then summed to yield a global PSQI score, which has a range of 0-21; higher scores indicate worse sleep quality (Buysse et al. 1989) . This tool has shown in its English version acceptable measures of internal homogeneity, consistency, and validity were obtained. A global PSQI score greater than 5 yielded a diagnostic sensitivity of 89.6% and specificity of 86.5% in distinguishing good and poor sleepers (Buysse et al. 1989) Tool that has been adapted in its Spanish version (Macias Fernandez and Royuela Rico 1996)

SECONDARY OUTCOMES:
Change in health-related quality of life , mesured with the Spanish version of EuroQol-5D Scale | Changes in baseline scores at 6 weeks (end of six sessions CBT - Intervention group), at 6 months (Intervention gruop & control group) and at 9 months (Intervention gruop & control group)
  Health-related quality of life (HRQoL) has been assessed using the EuroQol-5D Scale (EQ-5D) (EuroQol Group 1990) a self-applied scale that is quick and easy to administer, yielding a multidimensional description of general health as well as a numerical health profile. The scale is made up of two parts, the EQ-5D descriptive system, 5 dimensions (mobility, self- care, usual activities, pain/discomfort, and anxiety/de- pression), each with 3 levels of severity (value 1 = no problems, value 2 = some problems, value 3 = severe problems) and the visual analogue scale (EQ-VAS) (value 0 = worst and value 100 = best imaginable health status). This scale has been validated in Spain by Xavier Badia (Badia et al. 1999). For psychometric properties, the scale presented a test-retest reliability between 0.86 and 0.90 (van Agt et al. 1994) and a strong correlation with the SF-36 scale. The EQ-5D scale has also been shown to be valid for use with patients with schizophrenia (Prieto et al. 2004)

CONTACTS AND LOCATIONS:
Overall Officials: David Batalla-Martin, RN, MSc, Principal Investigator — Nou Barris Mental Health
Locations (1):
- Nou Barris Mental Health Center, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided